CLINICAL TRIAL: NCT01281995
Title: Effects of Systemically Administered Hydrocortisone on the Human Immunome in Healthy Volunteers
Brief Title: Effects of Systemically Administered Hydrocortisone on the Immune System in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110092; 11-H-0092
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08-30

CONDITIONS: Immunosuppression; Healthy; Healthy Subjects
Keywords: Biologic Samples; Hydrocortisone; Laboratory Research Specimens; Glucocorticoids; Immune Modulation; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Corticosteroids have been used to treat inflammation and immune system diseases for decades. However, despite their widespread use, there is little information on the specifics of how corticosteroids affect the immune system in humans. The Center for Human Immunology, Autoimmunity, and Inflammatory Diseases is interested in studying how the steroid hormone hydrocortisone affects the immune system in healthy volunteers, and in doing so to understand how hydrocortisone given at different doses works in treating many immune and inflammatory conditions.

Objectives:

- To evaluate the effects of hydrocortisone on the immune and inflammatory responses of healthy volunteers over the short and intermediate term (up to 28 days after administration).

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a full medical history and physical examination, and blood and urine tests. At this visit, participants will be separated into two groups, with each group scheduled to receive a different amount of hydrocortisone during the study visit.
* One week before the study visit, participants will provide a blood sample for baseline testing.
* Participants will be admitted for a 24-hour inpatient stay that will involve frequent blood draws. Between blood draws, participants will be able to work, watch TV, walk around, and so on, and will be provided with regular meals.
* Blood will be drawn 1 hour before the infusion of hydrocortisone. Participants will be divided into two further sets of groups with different blood draw schedules:
* Groups 1 (lower dose) and 2 (higher dose) will have blood draws 1, 4, 8, 12, and 24 hours after the hydrocortisone infusion.
* Groups 3 (lower dose) and 4 (higher dose) will have multiple blood draws over 24 hours, with timing based on data from the previous groups blood test results.
* Participants will provide additional blood samples 7 and 28 days after the in-patient visit....

DETAILED DESCRIPTION:
Corticosteroids have been in widespread therapeutic use as anti-inflammatory and immunomodulatory agents for decades, and there is a wealth of information on their immunosuppressive effects in animals and in human cells cultured in vitro. However, despite their ubiquitous clinical use, there is a paucity of information on the effects of corticosteroids administered to humans systemically, and no previous study has examined their effects on the human immunome.

Therefore the Center for Human Immunology, Autoimmunity, and Inflammatory Diseases proposes this protocol designed to obtain blood from healthy adult subjects at baseline, and then at various time points after administration of 250 mg and 50 mg of intravenous hydrocortisone. These samples will be used to perform a comprehensive and detailed analysis of the immune system in response to corticosteroid administration. To our knowledge, this protocol will be the first study to characterize the human cellular and molecular immune system parameters, or immunome, in healthy adult subjects after administration of corticosteroids. This information may be useful in understanding the mechanistic effects of this commonly prescribed class of medications in humans.

The primary objective is to perform laboratory studies to characterize the immune response in healthy adult volunteers after administration of moderate (250 mg) and low (50 mg) doses of the glucocorticoid hydrocortisone. Primary endpoint is the results of the research laboratory assessments. As samples will be stored indefinitely, the time frame for primary endpoint is indefinite.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteer (health status confirmed by History and Physical Exam and blood work)

Ages 18 years or older (no upper limit)

Must be willing to allow samples to undergo genetic studies

EXCLUSION CRITERIA:

Patients with diseases with an inflammatory or immune component

Patients who have irregular circadian rhythms, i.e. those who are blind or work night shifts

Patients with active infections requiring systemic antibiotic therapy

Use of immune modifying medications, i.e. NSAIDs (such as aspirin, ibuprofen (Advil, Motrin), naproxen (Aleve), celecoxib (Celebrex), ketorolac (Toradol) within the past month

Systemic fungal, viral, or mycobacterial infections

Persons who are alcoholic or abusers of illicit substances

Abnormal fasting glucose >100mg/dL

Female subjects may not be pregnant or lactating due to possible side effects of use of hydrocortisone in a non-benefit study

Liver function tests (AST, ALT, total bilirubin, alkaline phosphatase) above the normal laboratory reference range

Other contraindications to corticosteroids (i.e. gastrointestinal ulceration, Cushing s syndrome, congestive heart failure, uncontrolled hypertension, glaucoma, osteoporosis, or known hypersensitivity to corticosteroids)

Corticosteroid use within the last six months prior to enrollment, including topical, intra-articular or intramuscular injections, or inhaled administration

Prior use of systemically administered corticosteroids for >6 months duration

Use of azole medications or chronic opiates

Patients with psychiatric diagnoses or symptoms, to include hypomania, bipolar disorder, major depression, or dysthymia

Patients with a body mass index greater than 30

Subjects unable to comprehend the investigational nature of the study or those who are unable or unwilling to sign the consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01-21; Study Completion 2018-08-30

PRIMARY OUTCOMES:
Effects of hydrocortisone on the human immune

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Biancotto, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] HENCH PS, KENDALL EC, SLOCUMB CH, POLLEY HF. Effects of cortisone acetate and pituitary ACTH on rheumatoid arthritis, rheumatic fever and certain other conditions. Arch Intern Med (Chic). 1950 Apr;85(4):545-666. doi: 10.1001/archinte.1950.00230100002001. No abstract available. PMID 15411248
- [Background] Jaffe HL. THE INFLUENCE OF THE SUPRARENAL GLAND ON THE THYMUS : III. STIMULATION OF THE GROWTH OF THE THYMUS GLAND FOLLOWING DOUBLE SUPRARENALECTOMY IN YOUNG RATS. J Exp Med. 1924 Nov 30;40(6):753-9. doi: 10.1084/jem.40.6.753. PMID 19868956
- [Background] Ashwell JD, Lu FW, Vacchio MS. Glucocorticoids in T cell development and function*. Annu Rev Immunol. 2000;18:309-45. doi: 10.1146/annurev.immunol.18.1.309. PMID 10837061